CLINICAL TRIAL: NCT04767477
Title: Telerehabilitation and Face-to-face Rehabilitation on Tolerance to Exercise and Quality of Life of COVID-19 Survivors: a Study Protocol
Brief Title: Telerehabilitation and Face-to-face Rehabilitation on COVID-19 Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, BRUNA THAYS SANTANA DE ARAÚJO, physiotherapist, Universidade Federal de Pernambuco
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR and TR
Record Dates: First submitted 2020-12-21; First posted 2021-02-23 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-10

CONDITIONS: Covid19; Exercise Tolerance; Quality of Life; Lung Function; Fatigue Intensity
MeSH Terms: conditions — COVID-19; Fatigue | interventions — Telerehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Face-to-face rehabilitation and Telerehabilitation (Other): The Face-to-face rehabilitation and Telerehabilitation protocol will consist of flexibility exercises, aerobic and resistance training, with two sessions per week.
  Interventions: Other: Face-to-face rehabilitation; Other: Telerehabilitation

INTERVENTIONS:
Other: Face-to-face rehabilitation — Aerobic training will be performed with 60% to 80% of the maximum VO2 obtained through the CPET. The exercise will be performed on the treadmill, with a total time of 40 minutes, with 5 minutes of warm-up, 30 minutes of conditioning, 5 minutes of cooling down. Resistance training will be performed for upper and lower limbs and the load used in the exercises will be 60% of the maximum repetition test (1RM), with load progression every six sessions. The exercises are performed in three series of 12 repetitions.
Other: Telerehabilitation — The telerehabilitation protocol will consist of stretching the muscles of the upper and lower limbs and accessory muscles of breathing. The conditioning phase will consist of stationary walking, side running, jumping jump and stationary running, 3 times of 40 seconds with a 30-second passive rest interval between them. Resistance training will be applied to the muscles of the upper limbs and lower limbs, with specific exercises for each musculature, using elastic bands as resistance.

SUMMARY:
INTRODUCTION: As this is a new disease, the short- and long-term consequences for patients with COVID-19 are still unclear. The use of sedatives, as well as prolonged rest, can lead to musculoskeletal damage, including decreased muscle strength and physical function. Thus, rehabilitation after this disease is a key component in continuing patient care. OBJECTIVE: To verify the effects of face-to-face cardiac rehabilitation and telerehabilitation on tolerance to the maximum and submaximal exercise, lung function, fatigue intensity and quality of life of COVID-19 survivors. METHODS: This is a longitudinal, intervention study. Primary outcomes will be maximum and submaximal functional capacity, intensity and impact of fatigue, while secondary outcomes will be lung function and quality of life. EXPECTED RESULTS: This work will bring important information to the scientific community and health professionals, about the best forms of intervention and its repercussions on the surviving individuals of COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Adults of both genders;
* With a diagnosis of COVID-19 confirmed by a laboratory through RT-PCR means;
* Have to access to the internet and some device (smartphone, computer or notebook) that allows them to participate in the call centre.

Exclusion Criteria:

* Individuals with orthopaedic or neurological diseases;
* Individuals with difficulties in understanding and that present psychological changes that make it difficult or impossible to understand the information presented.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2021-03-28 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-09-10 (Actual)

PRIMARY OUTCOMES:
Maximum functional capacity | 12 weeks
  Evaluated by the cardiopulmonary exercise test by measuring the maximum oxygen consumption
Submaximal functional capacity | 12 weeks
  Evaluated by the six-minute walk test
Intensity and impact of fatigue | 12 weeks
  Evaluated by the Fatigue pictogram questionnaire, an ordinal scale composed of two questions graded in 5 captioned illustrations that assess the intensity (not at all tired, a little tired, moderately tired, very tired and extremely tired) and the impact of fatigue (I manage to do everything I normally do I do, I can do almost everything I usually do, I can do some of the things I usually do, I just do what I have to do and I can do very little).

SECONDARY OUTCOMES:
Spirometry | 12 weeks
  Number of patients with ventilatory disorder assessed by spirometry
Quality of life assessment: Short Form-36 questionnaire | 12 weeks
  In this questionnaire, a score of zero corresponds to the worst general health status and the one hundred best health status.

OTHER OUTCOMES:
Perception of clinical change | 12 weeks
  Evaluated by the Patient Global Impression of Change Scale which is a one-dimensional measure in which individuals can rate their associated improvement on a 7-item scale ranging from "1 = no changes" to "7 = much better".

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Federal de Pernambuco, Recife, Pernambuco, Brazil

IPD SHARING:
Plan to Share IPD: No